CLINICAL TRIAL: NCT00441766
Title: Safety and Efficacy of Oral AGN 203818 for the Relief of Irritable Bowel Syndrome Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to company decision after Part A. Part B was never conducted
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 203818-008
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2011-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- AGN 203818 3 mg (Experimental): Part A: AGN 203818 3mg capsule every 12 hours for 4 weeks
  Interventions: Drug: AGN 203818
- AGN 203818 20 mg (Experimental): Part A: AGN 203818 20mg capsule every 12 hours for 4 weeks
  Interventions: Drug: AGN 203818
- AGN 203818 60 mg (Experimental): Part A: AGN 203818 60mg capsule every 12 hours for 4 weeks
  Interventions: Drug: AGN 203818
- Placebo (Placebo Comparator): Part A: Placebo capsule every 12 hours for 4 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AGN 203818 — Part A: 3 mg AGN203818 capsule every 12 hours for 4 weeks
  Arms: AGN 203818 3 mg
Drug: AGN 203818 — Part A: 20 mg AGN203818 capsule every 12 hours for 4 weeks
  Arms: AGN 203818 20 mg
Drug: AGN 203818 — Part A: 60 mg AGN203818 capsule every 12 hours for 4 weeks
  Arms: AGN 203818 60 mg
Drug: placebo — Part A: placebo capsule every 12 hours for 4 weeks
  Arms: Placebo

SUMMARY:
This study will explore the safety and effectiveness of different doses of AGN 203818 in relieving Irritable Bowel Syndrome pain. The study is being conducted in 2 parts. Part A enrolled 213 pts dosed with either 3, 20, 60 mg AGN 203818 or placebo over 4 week treatment duration. Part B will enroll 320 pts and dose with either 60, 100, 160 mg BID AGN 203818 or placebo over 12 week treatment duration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Irritable Bowel Syndrome
* Moderate or severe IBS pain

Exclusion Criteria:

* Any other uncontrolled disease
* Pregnant or nursing females

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AGN 203818 3 mg: Part A: AGN 203818 3 mg capsule every 12 hours for 4 weeks
Period: Overall Study
Arm/Group | AGN 203818 60 mg | AGN 203818 20 mg | AGN 203818 3 mg | Placebo
Started | 53 | 53 | 53 | 54
Completed | 39 | 46 | 44 | 48
Not Completed | 14 | 7 | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN 203818 60 mg | AGN 203818 20 mg | AGN 203818 3 mg | Placebo | Total
Number analyzed (Participants) | 53 | 53 | 53 | 54 | 213
Age, Customized [Number; unit: participants]
  18 to 64 years | 48 | 48 | 50 | 54 | 200
  >=65 years | 5 | 5 | 3 | 0 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 53 | 54 | 213
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Highest-Average-Pain Score at Week 4
Description: Change from baseline in mean highest-average-pain score at Week 4. The mean highest-average-pain score was the average of the 7 highest daily-average-pain scores obtained over the 14 days prior to the Week 4 visit. Patients recorded their daily-average-pain on an 11-point scale (where 0 equals no pain and 10 equals worst pain imaginable). A negative number change from baseline represents a decrease in average pain (improvement).
Time Frame: Baseline, Week 4
Population: Modified Intent-To-Treat (m-ITT). The m-ITT population included all patients who started the study (randomized), who received the study medication and had at least one post-baseline mean highest-average-pain score.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | AGN 203818 60 mg | AGN 203818 20 mg | AGN 203818 3 mg | Placebo
Number analyzed (Participants) | 47 | 50 | 50 | 50
Scores on a Scale
  Baseline | 5.8 (1.18) | 5.7 (1.09) | 6.0 (1.48) | 6.0 (1.15)
  Change from Baseline at Week 4 | -2.3 (2.07) | -1.9 (1.81) | -1.7 (1.46) | -2.2 (2.15)

2. Secondary Outcome: Percentage of Patients Who Rated Their Condition as Improved on the Subject Global Impression of Change (SGIC) at Week 4
Description: Percentage of patients who rated their condition as improved on the SGIC at week 4. The SGIC score was assessed using a 7-point scale (score of 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse). Patients self-evaluated their overall change in symptoms (relief from symptoms of abdominal discomfort, pain, and altered bowel habits). An "improved" condition was defined as a score of 1, 2, or 3.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | AGN 203818 60 mg | AGN 203818 20 mg | AGN 203818 3 mg | Placebo
Number analyzed (Participants) | 47 | 50 | 50 | 50
Percentage of Patients | 76.1 | 73.5 | 85.7 | 77.5

3. Secondary Outcome: Percentage of Patients Who Experienced Adequate Relief of Irritable Bowel Syndrome (IBS) Pain (AR-IBS) at Week 4
Description: Percentage of patients who experienced AR-IBS at week 4. The AR-IBS is a self-evaluation by the patient of their perception of adequate relief of IBS pain over the last 7 days following treatment as compared to IBS pain before receiving treatment. Patients respond with either a "Yes" or "No", where "Yes" indicated adequate relief of pain and "No" indicated no relief from pain.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | AGN 203818 60 mg | AGN 203818 20 mg | AGN 203818 3 mg | Placebo
Number analyzed (Participants) | 47 | 50 | 50 | 50
Percentage of Patients | 60.9 | 58.0 | 61.2 | 67.3

4. Secondary Outcome: Change From Baseline in Frequency of Bowel Movements at Week 4 Using the Bristol Stool Scale (BSS)
Description: Change from baseline in the frequency of bowel movements per day using the BSS. The BSS categorizes stool based on the patient's description of its consistency. Patients are classified into 3 IBS subtypes according to their predominant stool patterns (C=constipation; D=diarrhea; M=mixed). A positive change from baseline in the IBS-C indicates improvement and a negative change from baseline in the IBS-D and IBS-M indicates improvement.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Bowel Movements (Stools) Per Day
Arm/Group | AGN 203818 60 mg | AGN 203818 20 mg | AGN 203818 3 mg | Placebo
Number analyzed (Participants) | 47 | 50 | 50 | 50
Bowel Movements (Stools) Per Day
  (IBS-C) Baseline | 0.9 (0.43) | 1.1 (0.47) | 1.0 (0.71) | 0.8 (0.57)
  (IBS-C) Change from Baseline at Week 4 | 0.1 (0.63) | 0.1 (0.72) | 0.0 (0.32) | 0.1 (0.50)
  (IBS-D) Baseline | 3.5 (1.59) | 3.6 (2.95) | 4.3 (2.48) | 3.4 (1.88)
  (IBS-D) Change from Baseline at Week 4 | -0.3 (1.10) | -0.8 (1.33) | -0.7 (1.09) | -0.4 (1.46)
  (IBS-M) Baseline | 1.3 (0.79) | 1.4 (0.78) | 2.7 (1.64) | 1.8 (1.41)
  (IBS-M) Change from Baseline at Week 4 | -0.2 (0.56) | -0.3 (0.68) | -0.1 (0.99) | 0.2 (0.86)

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs and AEs and is the total number of patients that were randomized (started the study) AND treated.
Arm/Group | AGN 203818 60 mg | AGN 203818 20 mg | AGN 203818 3 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 8/53 | 0/53 | 2/52 | 1/54
Other Adverse Events (participants affected / at risk) | 52/53 | 48/53 | 28/52 | 39/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN 203818 60 mg (N=53) | AGN 203818 20 mg (N=53) | AGN 203818 3 mg (N=52) | Placebo (N=54)
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Adjustment Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN 203818 60 mg (N=53) | AGN 203818 20 mg (N=53) | AGN 203818 3 mg (N=52) | Placebo (N=54)
Nausea (Gastrointestinal disorders) | 6 | 6 | 6 | 2
Abdominal Pain (Gastrointestinal disorders) | 5 | 4 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 3 | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 0 | 4
Flatulence (Gastrointestinal disorders) | 1 | 4 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 2 | 1
Fatigue (General disorders) | 4 | 5 | 2 | 3
Urinary tract infection (Infections and infestations) | 5 | 4 | 3 | 4
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1 | 3
Blood bilirubin decreased (Investigations) | 4 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 4 | 0 | 2 | 1
Reticulocyte count decreased (Investigations) | 0 | 3 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 1
Headache (Nervous system disorders) | 4 | 3 | 3 | 2
Somnolence (Nervous system disorders) | 3 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 5 | 1 | 3

LIMITATIONS AND CAVEATS:
Only Part A results are presented; Due to termination of the study, Part B was never conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.